CLINICAL TRIAL: NCT04176302
Title: Monitoring of Mobility of Parkinson's Patients for Therapeutic Purposes - Clinical Trial
Acronym: MoMoPa-EC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); European Regional Development Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: INV_PROC_A118; DTS17/00195 (Other Grant/Funding Number: Instituto de Salud Carlos III - European Regional Development Fund (ERDF))
Record Dates: First submitted 2019-11-18; First posted 2019-11-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Motor fluctuation; Parkinson; Accelerometer; Parkinson diary
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parkinson Holter (Active Comparator): The neurologists in the study will receive information from the Parkinson Holter (device being studied)
  Interventions: Device: Parkinson Holter
- Parkinson's diary (Active Comparator): The neurologists in the study will receive information from a motor fluctuations diary
  Interventions: Diagnostic Test: Motor fluctuations diary
- Traditional clinical practice (Placebo Comparator): The neurologists in the study will receive no additional information other than what is obtained during the visit
  Interventions: Other: Traditional clinical practice

INTERVENTIONS:
Device: Parkinson Holter — The neurologists will receive the wearable report (for medication adjustment, if any as per physician's criteria/judgement)
  Other Names: STAT-ON ® sensor
  Arms: Parkinson Holter
Diagnostic Test: Motor fluctuations diary — The neurologists will receive the patient's diary report (for medication adjustment, if any as per physician's criteria/judgement).
  Other Names: Parkinson's diary
  Arms: Parkinson's diary
Other: Traditional clinical practice — The neurologists will receive the patient & caregiver report at the time of the visit (for medication adjustment, if any as per physician's criteria/judgement).
  Other Names: Clinical interview
  Arms: Traditional clinical practice

SUMMARY:
When Parkinson Disease is mild, it responds well to treatment with drugs (L-Dopa and dopamine antagonists). However, as the disease progresses, the effect of the drugs diminishes and lasts for a shorter time (wearing-off), which require physicians to progressively increase and/or break up the dosage of dopamine drugs, to control symptoms over the course of the entire day. Despite this, most patients present motor fluctuations after 10 years. These fluctuations consist of changes between what are known as Off periods, when the medication does not produce an effect and mobility is hindered, and On periods when patients can move smoothly, with the medication producing its best effect.

The timeline of these motor fluctuations over the course of the day and also on different days is very valuable to precisely adjust the medication. Nevertheless, neurologists do not currently have detailed information on the timeline of the symptoms of their patients, which means that they have serious difficulties to obtain good results with the adjustment of medication. Currently, the neurologist's information on the time progression of the motor fluctuations is drawn from what the patient indicates in the office visit, or in the best case, from diaries that the patient fills out at home, periodically (e.g. every hour) noting the motor state (On or Off). Although the latter method is still the gold standard in research and in care, it has serious limitations, because patients often forget to record the information (especially when they are in Off), many do not recognize their motor states well, and few can maintain adherence to such a laborious system for more than a few days.

The Parkinson Holter (STAT-ON ®) is a wearable device, which objectively measures and records the motor fluctuations of the patients. It does not require intervention by the patient, and can, therefore, be used in daily life, long term if necessary. However, the concept that detailed knowledge of motor fluctuations of patients will lead to better control of the disease, thanks to optimisation of the therapeutic regimen, is still a hypothesis. To demonstrate or refute this hypothesis, we are now conducting a clinical trial, with this medical device, to study the clinical effectiveness in patients with moderate Parkinson's disease and motor fluctuations. This trial will show whether using the Parkinson Holter is better than the clinical interview used in traditional clinical practice (primary objective), and whether it is not inferior to the On-Off diary recorded by the patients at home (exploratory objective)

ELIGIBILITY:
Inclusion Criteria:

* Ideopathic Parkinson's Disease
* Disease in the moderate-severe phase (Hoehn & Yahr ≥ 2 en Off)
* Motor fluctuations (with at least 2h/day in Off)
* Agree to participate voluntarily and will sign a written consent form

Exclusion Criteria:

* Incapable of walking independently or H&Y=5
* Participating in another clinical trial
* Patients with acute intercurrent disease
* Psychiatric or cognitive disorders that prevent collaboration (MMSE <24)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Daily time in Off | 7 days
  Changes from baseline to last visit in daily hours in Off

SECONDARY OUTCOMES:
Number of clinical contacts | 6 months
  Number of patient visits and telephone controls to adjust medication
Patient's adherence to the MF measurement system | 7 days
  Total hour/days with information registered.
Number of therapeutic changes. | 6 months
  Number of therapeutic changes done to improve symptoms.
Motor complications | 6 months
  Changes from baseline to last visit in motor complications, assessed by means of Unified Parkinson's Disease Rating Scale - part IV
Daily time in On | 7 days
  Changes from baseline to last visit in daily hours in On
Change of presence and severity of freezing of gait episodes | 7 days
  Changes from baseline to last visit in the number and severity of freezing of gait episodes, assessed by means of Freezing of Gait Questionnaire
Reported quality of life | 1 month
  Changes from baseline to last visit in quality of life, assessed by menas of Parkinson's Disease Questionnaire-39
Activities of Daily Living | 6 months
  Changes from baseline to last visit in dependence for Activities of Daily Living assessed by means of Unified Parkinson's Disease Rating Scale - part II
User satisfaction: Quebec User Evaluation of Satisfaction with assistive Technology | 7 days
  Physician and patient satisfaction with the Parkinson Holter will be assessed by means of the Quebec User Evaluation of Satisfaction with assistive Technology (QUEST)
System usability: System Usability Scale | 7 days
  Usability of the system will be assessed by System Usability Scale (SUS)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Rodríguez-Molinero, PhD/MD, Study Director — Consorci Sanitari de l'Alt Penedès i Garraf
Locations (43):
- Spain (43):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital General de l'Hospitalet. CS Integral, L'Hospitalet de Llobregat, Barcelona
  - Consorci Sanitari del Maresme. Hospital de Mataró, Mataró, Barcelona
  - Hospital Universitari Mútua Terrassa, Terrassa, Barcelona
  - Consorci Sanitari de l'Alt Penedès i Garraf, Vilafranca del Penedès, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital General La Mancha-Centro, Alcázar de San Juan, Alcázar de San Juan, Ciudad Real
  - Hospital Universitario Lucus Augustí, Lugo, Galicia
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Guipúzkoa
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario del Henares, Madrid, Madrid
  - Hospital Universitario La Princesa, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Majadahonda, Madrid
  - Hospital Univesitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital General de Elche, Alicante
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Moisès Broggi - CS Integral, Barcelona
  - Hospital Sanitas CIMA, Barcelona
  - Terapia Integral UParkinson, SL, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitari dr. Josep Trueta, Girona
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Moraleja, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes
  - Hospital General Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Virgen del Rocío, Seville
  - Consorci Sanitari de Terrassa, Terrassa
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital de Llíria, Valencia
  - Hospital Royo de Vilanova, Zaragoza

REFERENCES:
- [Result] Rodriguez-Molinero A, Perez-Lopez C, Caballol N, Buongiorno M, Avila Rivera MA, Lopez Ariztegui N, Lopez-Manzanares L, Hernandez-Vara J, Bayes-Rusinol A, Gironell Carrero A, Alvarez Sauco M, Franquet Gomez E, Perez-Martinez DA, Escalante Arroyo S, Marti-Martinez S, Mir P, Salom Juan JM, Martinez-Castrillo JC, Tebe C; MoMoPa-EC Research Group. Parkinson's disease medication adjustments based on wearable device information compared to other methods: randomized clinical trial. NPJ Parkinsons Dis. 2025 Aug 20;11(1):249. doi: 10.1038/s41531-025-00977-2. PMID 40835832
- [Derived] Perez-Lopez C, Hernandez-Vara J, Caballol N, Bayes A, Buongiorno M, Lopez-Ariztegui N, Gironell A, Lopez-Sanchez J, Martinez-Castrillo JC, Sauco M A, Lopez-Manzanares L, Escalante-Arroyo S, Perez-Martinez DA, Rodriguez-Molinero A; MoMoPa-EC Research Group. Comparison of the Results of a Parkinson's Holter Monitor With Patient Diaries, in Real Conditions of Use: A Sub-analysis of the MoMoPa-EC Clinical Trial. Front Neurol. 2022 May 16;13:835249. doi: 10.3389/fneur.2022.835249. eCollection 2022. PMID 35651347
- [Derived] Rodriguez-Molinero A, Hernandez-Vara J, Minarro A, Perez-Lopez C, Bayes-Rusinol A, Martinez-Castrillo JC, Perez-Martinez DA; Monitoring Parkinson's patients Mobility for therapeutic purposes research group. Multicentre, randomised, single-blind, parallel group trial to compare the effectiveness of a Holter for Parkinson's symptoms against other clinical monitoring methods: study protocol. BMJ Open. 2021 Jul 19;11(7):e045272. doi: 10.1136/bmjopen-2020-045272. PMID 34281918